CLINICAL TRIAL: NCT02282423
Title: PGC-1 & Muscle Mitochondrial Dysfunction in Diabetes
Acronym: PGC-1
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI job change
Sponsor: Mayo Clinic (Other)
Collaborators: Arizona State University (Other)
Responsible Party: Principal Investigator, Lawrence Mandarino, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 13-006411
Record Dates: First submitted 2014-10-29; First posted 2014-11-04 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus; Obesity | interventions — Glucose Tolerance Test; Glucose Clamp Technique

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Lean Controls (Experimental): Lean controls will have BMI of 25 or less, gender specific normal body fat, and not be taking any medication that affects glucose metabolism.
  Interventions include OGTT, Clamp, VO2 Max, Exercise Test and Muscle Biopsy
  Interventions: Behavioral: Pre-study dietary and exercise instruction.; Procedure: Screening examination and oral glucose tolerance test; Procedure: Euglycemic clamp; Procedure: VO2max.; Behavioral: Acute exercise bout; Procedure: Percutaneous needle muscle biopsies
- Obese, Non-diabetic (Experimental): Obese nondiabetics will have a BMI between 30-50 and not be taking any medication that affects glucose metabolism.
  Interventions include OGTT, Clamp, VO2 Max, Exercise Test and Muscle Biopsy
  Interventions: Behavioral: Pre-study dietary and exercise instruction.; Procedure: Screening examination and oral glucose tolerance test; Procedure: Euglycemic clamp; Procedure: VO2max.; Behavioral: Acute exercise bout; Procedure: Percutaneous needle muscle biopsies
- Diabetic (Experimental): Diabetic patients will have a BMI between 30-50. We will recruit patients with mild or newly diagnosed type 2 diabetes who are treated with diet, sulfonylureas, or other drugs working through enhanced insulin secretion. Patients taking metformin or TZDs will not be recruited due to the effects of those drugs on insulin action.
  Interventions include OGTT, Clamp, VO2 Max, Exercise Test and Muscle Biopsy
  Interventions: Behavioral: Pre-study dietary and exercise instruction.; Procedure: Screening examination and oral glucose tolerance test; Procedure: Euglycemic clamp; Procedure: VO2max.; Behavioral: Acute exercise bout; Procedure: Percutaneous needle muscle biopsies
- Non-diabetic (Experimental): Patients will be nondiabetic, although we will include patients with impaired glucose tolerance. Patients will meet criteria for treatment with fibrates to lower plasma triglyceride concentrations (triglyceride>300 mg/dl for nondiabetics, 250 mg/dl for patients with impaired glucose tolerance). We will aim at recruiting equal numbers of men and women. All participants will be between the ages of 30 and 59. Patients will have a BMI of 25-50 and not be taking any other medication that affects glucose metabolism. All participants will be sedentary (not reporting more than 10 minutes per day of light to vigorous leisure time physical activity.
  Interventions include OGTT, Clamp, VO2 Max, Exercise Test and Muscle Biopsy
  Interventions: Behavioral: Pre-study dietary and exercise instruction.; Procedure: Screening examination and oral glucose tolerance test; Procedure: Euglycemic clamp; Procedure: VO2max.; Behavioral: Acute exercise bout; Procedure: Percutaneous needle muscle biopsies

INTERVENTIONS:
Behavioral: Pre-study dietary and exercise instruction. — All subjects will be instructed to continue their normal diet during the three days prior to study, to not consume alcohol the day before study, and to not engage in exercise for 48 hours before all studies.
Procedure: Screening examination and oral glucose tolerance test — All subjects will have screening exam and OGTT at the Clinical Studies Infusion Unit at Mayo Clinic in Arizona at 7-8 am after having eaten nothing after 10 PM the night before, and have a screening examination and 75 g OGTT, as described
  Other Names: OGTT
Procedure: Euglycemic clamp — On a separate day, subjects will have a two-hour euglycemic clamp ((80 mU insulin/(m2.min)) at the Clinical Studies Unit at Mayo Clinic Arizona at 7-8 am after an overnight fast. A muscle biopsy will be taken before the insulin infusion, to serve as the resting biopsy (3). Biopsy specimens (150-300 mg) will be frozen immediately in liquid nitrogen and stored in liquid nitrogen until they are processed
Procedure: VO2max. — VO2max.
Behavioral: Acute exercise bout — The single acute exercise bout will be performed as described (3). It consists of 4 sets of 12 min each (8 min @ 70% VO2max, 2 min @ 90%, 2 min rest, repeat X 4). Biopsies are taken 30 min and 24 hr after end of exercise. Resting biopsies are taken on the glucose clamp day
Procedure: Percutaneous needle muscle biopsies — Skeletal muscle biopsies, blotted free from blood, are frozen within 30 seconds in liquid nitrogen, and stored in liquid nitrogen until processing. We routinely obtain 150-300 mg muscle (wet weight), which is more than sufficient for the analyses proposed, with some muscle remaining for any additional validation assays that may arise during the course of the research. Muscle will be processed either for isolation of mRNA/microRNA or protein, as described (2, 3, 12).

SUMMARY:
The goal of this study is to understand how and why insulin resistant individuals respond differently to exercise as compared with insulin sensitive individuals at the skeletal muscle and gene expression level.

DETAILED DESCRIPTION:
The goal of this study is to understand how and why insulin resistant individuals respond differently to exercise as compared with insulin sensitive individuals at the skeletal muscle and gene expression level. The study has four aims including testing if MZF1, NFKB1, RELA, SP1/KLF and EGRI expression responses are outside of the normal range in insulin resistant individuals and how insulin resistance changes the cell biosynthesis process/ post translational modifications. It also aims to define the response of MiRNAs in healthy and insulin resistant individuals and determine if treatment with Gemfibrozil inhibits transcription processes.

ELIGIBILITY:
Inclusion Criteria: Aims1-3

1. Age 30-59
2. BMI: Lean, BMI less than or equal to 25; Obese, BMI between 30-40; type 2 diabetic, BMI between 30-40.
3. Subjects must be able to communicate meaningfully with the investigator and must be legally competent to provide written informed consent.
4. Subjects may be of either sex with age as described in each protocol. Female subjects must be non-lactating and will be eligible only if they have a negative pregnancy test throughout the study period.
5. Subjects must range in age as described in each specific protocol.
6. Subjects must have the following laboratory values:

   * Hematocrit ≥ 35 vol%
   * Serum creatinine ≤ 1.6 mg/dl
   * AST (SGOT) < 2 times upper limit of normal
   * ALT (SGPT) < 2 times upper limit of normal
   * Alkaline phosphatase < 2 times upper limit of normal
   * Triglycerides < 150 mg/dl (except for Aim 4).

Aim 4

1. Age 30-59
2. BMI: Lean, BMI less than or equal to 25; Obese, BMI between 30-40.
3. Patients may have normal or impaired glucose tolerance.
4. Subjects must be able to communicate meaningfully with the investigator and must be legally competent to provide written informed consent.
5. Subjects may be of either sex with age as described in each protocol. Female subjects must be non-lactating and will be eligible only if they have a negative pregnancy test throughout the study period.
6. Subjects must have the following laboratory values:

   * Hematocrit ≥ 35 vol%
   * Serum creatinine ≤ 1.6 mg/dl
   * AST (SGOT) < 2 times upper limit of normal
   * ALT (SGPT) < 2 times upper limit of normal
   * Alkaline phosphatase < 2 times upper limit of normal
   * Triglycerides > 300 mg/dl for nondiabetics, > 250 mg/dl for impaired glucose tolerance.

Exclusion Criteria:

1. Subjects must not be receiving any of the following medications: thiazide or furosemide diuretics, beta-blockers, or other chronic medications with known adverse effects on glucose tolerance levels unless the patient has been on a stable dose of such agents for the past three months before entry into the study. Subjects may be taking a stable dose of estrogens or other hormonal replacement therapy, if the subject has been on these agents for the prior three months. Subjects taking systemic glucocorticoids are excluded. Patients with type 2 diabetes will be excluded if they are taking metformin or thiazolidinediones, but may be taking sulfonylureas or other medications known to work through effects on insulin secretion.
2. Subjects receiving Gemfibrozil must not also be receiving a statin.
3. Subjects with a history of clinically significant heart disease (New York Heart Classification greater than grade II; more than non-specific ST-T wave changes on the EKG), peripheral vascular disease (history of claudication), or pulmonary disease (dyspnea on exertion of one flight or less; abnormal breath sounds on auscultation) will not be studied.
4. Recent systemic or pulmonary embolus, untreated high-risk proliferative retinopathy, recent retinal hemorrhage, uncontrolled hypertension, systolic BP>180, diastolic BP>105, autonomic neuropathy, resting heart rate >100, electrolyte abnormalities.

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2014-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Transcription Factor Response to Exercise | 4-6 weeks
  To determine whether expression of the transcription factor MZF1 is induced by exercise to a greater degree in control patients than in those with type 2 diabetes mellitus. MZF1 expression will be determined using quantitative rt-PCR analysis on RNA isolated from muscle biopsies taken from the patients. An repeated measures analysis of variance will be performed on the PCR data, for the three groups (lean, obese, type 2 diabetic), with the difference between the lean and diabetic groups being the primary measure. A P value of 0.05 will be considered significant.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence J. Mandarino, Ph.D., Principal Investigator — Mayo Clinic; Lori Roust, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Scottsdale, Arizona, United States